CLINICAL TRIAL: NCT05562700
Title: Assessment of Return to Work and Functional Results of French Military Personnel After Ankle Ligamentoplasty
Acronym: LITCHEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PPRC14; 2022-A01577-36 (Other: IDRCB)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Ankle Sprains
Keywords: Ligamentoplasty
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: On-line questionnaire — It is a self-administered questionnaire (20 minutes) with several subparts:
  * Socio-demographic questions: age, height, weight, smoking status, etc.
  * Care: date of accident, initial treatment, duration of symptoms, complications, return to work, return to sport, recovery of skills, etc.
  * Functional results

SUMMARY:
In the general population, ankle sprains are one of the most common injuries, accounting for approximately 20% of all sports injuries and the most frequent reason for trauma consultation (4 to 7% of admissions to emergency departments in France).

The most frequent complication after an episode of ankle sprain is the development of chronic ankle instability (5 to 40% of the patients). Chronic ankle instability is defined by a history of at least one significant ankle sprain with subsequent perception of an abnormal ankle by the patient, associated with various symptoms including: recurrent sprains, repeated episodes of ankle "slippage", pain, episodes of swelling, difficulty and apprehension when walking on uneven surfaces with a decrease in the functional capacity of the ankle or restriction of activity.

In the military population, ankle sprains account for 18.60% of on-duty injuries, and epidemiologic studies report an incidence of 45.14 to 58.40 sprains per 1,000 person-years.

A 2019 study in a population of French military paratroopers found a prevalence of chronic ankle instability of 43.1% after an ankle sprain.

Chronic ankle instability leads to a loss of operational skills in French soldiers, since it results in a score of 4 for the letter "I" (pelvic girdle and lower limbs) in the SIGYCOP military medical profile. The treatment of chronic ankle instability after failure of rehabilitation consists in ligamentoplasty, conservative or not, in order to restore an external ligament plane and stabilize the ankle. For open techniques, the median time to return to sport after ligamentoplasty is 4.7 months. In the series by Lee et al, which studied more specifically the return to sport in high-level athletes, 83.3% of athletes had returned to competitive sport at 4 months and 100% at 8 months. Management of chronic ankle instability by ligamentoplasty may allow the soldier to regain his operational ability (SIGYCOP score I=2).

ELIGIBILITY:
Inclusion Criteria:

* Military personnel,
* Primary ankle ligamentoplasty surgery between January 2015 and December 2021,
* Sufficient French language reading/writing level (elementary school level).

Exclusion Criteria:

* Ankle ligament surgery after a first failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of military personnel who have undergone primary ankle ligamentoplasty surgery between January 2015 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who returned to their previous job six months after ankle ligamentoplasty surgery | Through study completion (12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Percy, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided